CLINICAL TRIAL: NCT00988520
Title: Study of Efficacy, Pharmacokinetics and Safety of Continuous Intravenous Infusion of Org 9426 Following a Single Intubating Dose in Adult Patients Undergoing Operation Under Sevoflurane or Propofol Anesthesia.
Brief Title: Study of Efficacy, Pharmacokinetics and Safety of Continuous Intravenous Infusion of Org 9426 (Study P05977)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P05977; 71103
Record Dates: First submitted 2009-10-01; First posted 2009-10-02 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Anesthesia
Keywords: Neuromuscular Blocking Agents
MeSH Terms: interventions — Rocuronium; Sevoflurane; Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 0.6 mg/kg intubation dose under sevoflurane (Experimental)
  Interventions: Drug: Rocuronium bromide; Drug: Sevoflurane
- 0.9 mg/kg intubation dose under sevoflurane (Experimental)
  Interventions: Drug: Rocuronium bromide; Drug: Sevoflurane
- continuous dose following 0.6 mg/kg intubation dose + propofol (Experimental)
  Interventions: Drug: Rocuronium bromide; Drug: Propofol
- continuous dose following 0.9 mg/kg intubation dose + propofol (Experimental)
  Interventions: Drug: Rocuronium bromide; Drug: Propofol

INTERVENTIONS:
Drug: Rocuronium bromide — Continuous intravenous infusion initiated at 7 μg/kg/min and adjusted to maintain muscle relaxation
  Other Names: SCH 900085
Drug: Rocuronium bromide — Intubation dose of 0.6 mg/kg injection
  Other Names: SCH 900085
  Arms: 0.6 mg/kg intubation dose under sevoflurane; continuous dose following 0.6 mg/kg intubation dose + propofol
Drug: Rocuronium bromide — Intubation dose of 0.9 mg/kg injection
  Other Names: SCH 900085
  Arms: 0.9 mg/kg intubation dose under sevoflurane; continuous dose following 0.9 mg/kg intubation dose + propofol
Drug: Sevoflurane — 0.5-2.0% intravenous maintenance anesthesia
  Other Names: Sevofrane
  Arms: 0.6 mg/kg intubation dose under sevoflurane; 0.9 mg/kg intubation dose under sevoflurane
Drug: Propofol — 4010 mg/kg/hr intravenous maintenance anesthesia
  Other Names: Diprivan
  Arms: continuous dose following 0.6 mg/kg intubation dose + propofol; continuous dose following 0.9 mg/kg intubation dose + propofol

SUMMARY:
The purpose of this study is to compare the infusion rate of Org 9426 following intubating dose of Org 9426 0.6 mg/kg or 0.9 mg/kg in adult surgical patients.

ELIGIBILITY:
Inclusion Criteria:

* Subjects at least 20 but under 65 years of age.
* Subjects of asa class 1, 2 or 3 for general elective surgery.
* Subjects who are not considered to be pregnant.
* Subjects scheduled for elective surgery under sevoflurane or propofol anesthesia, with anticipated duration of surgery of 2-5 hours.
* Subjects with normal laboratory values for serum electrolytes (Na+, K+, Cl-), BUN, creatinine, total bilirubin, ALP, ALAT and ASAT as judged by the investigator or the sub-investigator.
* Subjects who received an explanation of the trial and agreed informed consent in writing to participate in the trial in advance.

Exclusion Criteria:

* Subjects with renal dysfunction as a complication or in the history.
* Subjects with serum creatinine level greater than 1.6 mg/dL.
* Subjects with severe hepatic dysfunction as a complication or in the history.
* Subjects with known significant metabolic or neuromuscular disorders.
* Subjects with showing dyspnea, airway obstruction or bronchial asthma.
* Subjects with a history of hypersensitivity to pancuronium bromide, vecuronium bromide or bromine.
* Subjects with atopic diseases.
* Subjects who have developed any systemic allergic symptoms related to drugs or general anesthesia.
* Subjects receiving antihistamines and antiallergic agents for 1 month or more.
* Subjects receiving any of the following drugs known to affect on the action of neuromuscular blocking agents on surgery day: calcium antagonists; anticonvulsants; aminoglycoside antibiotics; polypeptide antibiotics; or metronidazole.
* Subjects under hypothermic anesthesia.
* Subjects who participated as research subjects in another trial within the last 6 months or is now participating in other trials.
* Other subjects judged to be ineligible as subjects in this trial by the discretion of the investigator or sub-investigator.

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2003-05; Primary Completion 2003-09 (Actual); Study Completion 2003-09 (Actual)

PRIMARY OUTCOMES:
Infusion rate following intubation doses of 0.6 mg/kg or 0.9 mg/kg | 90 minutes after start of continuous infusion